## **Participant Informed Consent for Clinical Research**

**Study title for participants:** Imaging Study of 18F-FAC PET Scans to Assess Standard Treatment in People with Pancreatic Cancer

Official study title for internet search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: 18F-FAC PET Imaging to Quantify Gemcitabine Tumor Drug Uptake and Biodistribution in Pancreatic Cancer Patients

Lead Researcher: Heiko Schöder, MD (646-634-2751)

If you are the legally authorized representative (LAR) of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to the study participant.

### **Overview and Key Information**

### Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

You are being asked to take part in this study because you have pancreatic ductal adenocarcinoma (PDAC) and you may receive chemotherapy, which is the standard treatment for your cancer.

It can be difficult to know whether this treatment is being absorbed by your tumor(s), which makes it hard to tell whether the chemotherapy is effectively treating your cancer. The study researchers think that performing a PET (positron emission tomography) scan with an experimental imaging tracer called 18F-FAC may show how much of the chemotherapy drug is taken up by your cancer and other organs. The 18F-FAC gives off a small amount of radiation, which makes it easy to see on PET scans. And although 18F-FAC and the chemotherapy drug are different drugs, they are distributed through the body and absorbed in similar ways, so the 18F-FAC that "lights up" on the PET scan can show how much of the chemotherapy drug may reach your tumor, which is needed to destroy your cancer cells.

The US Food and Drug Administration (FDA) has not approved 18F-FAC PET imaging to assess the effectiveness of treatment for PDAC or any other disease. The use of 18F-FAC PET imaging in this study is considered investigational, and the results of this imaging procedure will not be used to guide or change the usual care for your cancer.

## Taking part in this study is your choice.

You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered.

# What is the usual approach to treating PDAC?



People who are not in a research study are usually treated with chemotherapy, and they may have imaging procedures (MRI/PET/CT scans) during the standard treatment for their cancer. However, they do not have research imaging procedures before treatment.

## What are my other choices if I decide not to take part in this study?

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available
- You may choose not to be treated for cancer
- You may choose not to be treated for cancer, but to receive comfort care to help relieve your symptoms

## What will happen if I decide to take part in this study?

If you decide to take part in this study, before you begin to receive the standard treatment for your cancer we will give you an intravenous (IV) injection of 18F-FAC and perform a PET scan.

We will draw two blood samples (each about 3 ml) within the first 5 minutes after the 18F-FAC injection.

During or following chemotherapy or radiation therapy, you will be given an opportunity to receive an optional second PET scan to study changes in drug uptake and distribution.

We will monitor your condition after you receive the injection and during the scanning procedure, and you will be able to leave the clinic after the scan has been completed. The study doctor will contact you by phone within one to three business days after the completed scan, to ask whether you are having any side effects from the injection of the tracer.

The study team will continue to follow your condition throughout your life during your regularly scheduled clinic visits.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### **Risks**

We want to make sure that you know about a few key risks right now. We will also give you more information in the *What risks can I expect from taking part in this study?* section of this consent form.

If you choose to take part in this study, there is a risk that the 18F-FAC PET scan may not show whether/how much of the standard chemotherapy may reach your cancer cells.

There is also small risk that you could have side effects from the 18F-FAC PET scan. These side effects may be different than you would have with standard PET imaging.

The imaging agent has been studied in healthy volunteers at another hospital in the US, and no side effects have been reported to date. There may be some risks that the study doctors do not yet know about.

**Possible risks of collecting a blood sample:** We do not expect you to experience any physical injuries while you are participating in this study. You may have slight discomfort and/or bruising at the



place on your arm where the needle is inserted to collect your blood. Rarely, an infection may occur at this site.

#### **Benefits**

You will not benefit directly from participating in this study. What we learn from this study may help other people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest
- You do not follow the study rules
- For participants who are able to have children: You become pregnant while you are in the study
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), US Food and Drug Administration (FDA), or the study sponsor, Memorial Sloan Kettering Cancer Center (MSK). The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

## What is the purpose of this study?

The purpose of this study is to find out whether a pre-treatment PET scan using the experimental imaging tracer 18F-FAC can show how much of the standard chemotherapy for PDAC may be taken up by your cancer.

18F-FAC gives off a small amount of radiation, which makes it easy to see on PET scans. Because this experimental imaging tracer and the chemotherapy are distributed through the body and absorbed in very similar ways, an 18F-FAC PET scan may show whether the chemotherapy will be absorbed by your tumor(s), which is needed to destroy your cancer cells.

The 18F-FAC used in this study will be provided by the study sponsor, Memorial Sloan Kettering Cancer Center.



About 30 people will take part in this study at Memorial Sloan Kettering Cancer Center (MSK).

### What are the study groups?

All study participants will have an 18F-FAC PET scan before starting standard chemotherapy for PDAC. All study participants will also receive two blood draws after the 18F-FAC injection. Participants will be given an opportunity to receive an optional second PET scan during or after chemotherapy or radiation therapy.

## What extra tests and procedures will I have if I take part in this study?

#### Before you begin the main part of the study:

The study doctor will review your medical records and the results of your exams, tests, and procedures to see if it is safe for you to take part in the study. This first part of the study is called screening. All the screening exams, tests, and procedures are part of the usual care that you would have if you were not in a study.

#### **During the study:**

Within 4 weeks before you start chemotherapy for PDAC, you will come to the clinic to receive an intravenous (IV) injection of the imaging tracer 18F-FAC. Then you will have a PET scan. The imaging procedure will last about 1 hour.

Two blood samples will be collected within 5 minutes after the 18F-FAC injection for research testing to find out the stability of the parent [18F]-FAC radiotracer compound for further refinement of the kinetic modeling analysis.

About one tablespoon of blood will be collected from a vein in your arm.

During or following chemotherapy or radiation therapy, you will be given an opportunity to receive an optional second PET scan to study changes in drug uptake and distribution.

We will monitor your condition after you receive the injection and during the scanning procedure, and you will be able to leave the clinic after the scan has been completed. A study doctor will contact you by phone within one to three business days after the completed scan, to ask whether you are having any side effects from the injection of the tracer.

#### Exams, Tests and/or Procedures

After the PET scans and blood draws described above, you will not have any additional tests or procedures done only for research purposes.

#### Follow-up:

The study team will continue to follow your condition throughout your life during your regularly scheduled clinic visits.

#### Will I receive the results of my research tests?

You will receive the results of any tests done only for research purposes during this study.

# What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:



Page 4 of 13

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office
- You may be asked sensitive or private questions that you do not usually discuss

The radiotracer may cause an allergic reaction. Symptoms of allergic reactions include hives or skin rash, swelling of the face, difficulty breathing, nausea, vomiting, or low blood pressure (causing you to feel faint). Allergic reactions may be mild or severe. Rarely, these reactions may lead to death.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Important information about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may be mild. Others may be very serious and may even result in death.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor may be able to treat some side effects.

Because the radiotracer used in this study has not been tested in large numbers of people, we may not know all the side effects that may occur. If important new side effects are found during this study, the study doctor will discuss them with you.

**Possible risks of radiation-based diagnostic imaging:** You will be exposed to low amounts of radiation from the radiotracer and the imaging procedures performed during this study. The PET scans provide detailed pictures of the inside of the body, like an MRI (magnetic resonance imaging) scan, but using radiation, like an X-ray. Every day, people are exposed to low levels of radiation that comes from the sun and the environment. Scientists think that exposure to too much radiation can be harmful. The amounts of radiation associated with the scan(s) included in this study are comparable to those from standard-of-care imaging procedures. Each year, many thousands of patients routinely undergo similar diagnostic procedures and receive comparable radiation doses with no short- or long-term adverse effects.

**Reproductive risks**: You should not get pregnant, breastfeed, father a baby, or donate sperm while you are in this study. The imaging agent/procedure used in this study could be very damaging to an unborn baby. Check with the study doctor about what types of birth control or pregnancy prevention to use while you are in this study.

Let the study doctor know about any questions you may have about possible side effects. You can ask the study doctor questions about side effects at any time.

**Possible risks of collecting a blood sample:** We do not expect you to experience any physical injuries while you are participating in this study. You may have slight discomfort and/or bruising at the place on your arm where the needle is inserted to collect your blood. Rarely, an infection may occur at this site.



### What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments
- Tell the study doctor about:
  - All medications and any supplements you are taking
  - o Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - o Whether you have been or are currently in another research study

### Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Center. There are no known investigator and/or institutional conflicts of interest for this study.

## What are the costs of taking part in this study?

You will not have to pay for the 18F-FAC imaging tracer, research blood draws, or for the research PET scans.

You and/or your health plan/insurance company will have to pay for all the other costs of treating your cancer while you are in this study. These charges include the costs of insurance co-pays and deductibles, as well as tests, procedures, or drugs that you get during the study to monitor your safety, and to prevent or manage any side effects.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this clinical trial. Also find out if you need approval from your health plan before you can take part in this study.

The study doctor or nurse can help you find the right person to talk to if you are not sure which costs will be billed to you or your insurance provider.

## Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company.

If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.



### Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.

In the future, your information (data) may be de-identified, which means that your data and/or biospecimens will be assigned a unique code, and the list that links the code to your name will be stored separately from your biospecimens and data. Your de-identified information may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK, and may be stored in public databases related to research. All requests for data sharing will be reviewed by the study sponsor, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or Social Security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.

## Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.

#### **Optional Studies:**



# Memorial Sloan Kettering Cancer Center IRB Number: 21-442 A(5) Approval date: 02-Aug-2023

This part of the consent form describes an optional study that you can choose to take part in. You will not get health benefits from this study. The doctors leading this research hope that the results of this study will help other people with cancer in the future.

The results of this study will be added to your medical records, and you and/or your study doctor will be informed of the test results.

You will not be billed for this optional study. You can still take part in the main study even if you do not participate in the optional study. If you sign up for but cannot complete the optional study for any reason, you can still take part in the main study.

#### Optional imaging study: Research scan or procedure

If you choose to take part in this optional imaging study, you will receive an additional dose of the 18F-FAC PET tracer as well as an additional PET scan to study changes in drug uptake and distribution. The scan will be done during or following chemotherapy or radiation therapy.

The scan will be used only for research, and not to guide your medical care. You will receive the results of any tests done only for research purposes during this study.

You will be exposed to low amounts of radiation from the imaging procedures performed during this study. The PET scans provide detailed pictures of the inside of the body, like an MRI (magnetic resonance imaging) scan, but using radiation, like an X-ray. Every day, people are exposed to low levels of radiation that comes from the sun and the environment. Scientists think that exposure to too much radiation can be harmful.

The amounts of radiation associated with the scan(s) included in this study are comparable to those from standard-of-care imaging procedures. Each year, many thousands of patients routinely undergo similar diagnostic procedures and receive comparable radiation doses with no short- or long-term adverse effects.

Contrast materials, also called contrast agents or contrast media, are injected into a vein in the arm to improve the pictures produced by PET scans and MRI scans. Contrast materials are generally very safe, but adverse reactions ranging from mild to severe may occur. Serious allergic reactions or other reactions are rare. A small percentage of patients may develop a delayed allergic reaction, with a rash that can occur hours to days after the injection of the contrast agent. Most of these rashes are mild, but severe rashes may require medication; please discuss any reactions with the study doctor.

Please check Yes or No. Your medical care will not be affected, no matter what you decide to do.

I agree to have the experimental 18F-FAC PET.

☐ Yes ☐ No



# Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

Imaging Study of 18F-FAC PET Scans to Assess Standard Treatment in People with Pancreatic Cancer

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

# 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- Any health information or clinical data associated with your biospecimens, if the information or data could be reasonably used to identify you. This information or data will be shared only if you have agreed to it by signing this informed consent document.
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

# 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigators: Heiko Schöder, MD; John Humm, Ph.D.; and Kenneth Yu, MD
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



# 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study drug.
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)
- Other qualified researchers, approved by Memorial Sloan Kettering Cancer Center, who may receive individual research results that do not identify you.

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

# 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

# 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the study may be analyzed for many years, and it is not possible to know when this analysis will be completed.



## 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be able to participate in this research study. However, if you do not sign, it will not affect your ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to the parts of your medical record that are unrelated to this study at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

#### **Notice concerning HIV-related information**

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your rights.



Participant Informed Consent/Research Authorization for Clinical Research Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information, including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

| Consenting professional's | Date: |
|---|---|
| signature | |
| Consenting professional's name (Print) | |
| Participant's (or Legally Authorized Representative's [LAR's)]) statement | |
| I have read this form that describes the clinical research study. I have also talked it over to my satisfaction with the consenting professional. By signing below, I agree to the following: (1) to voluntarily participate in | |
| this clinical research study; (2) to authorize the use and disclosure of my/the participant's protected health | |

Consenting professional must personally sign and date

of this consent form.

Participant/LAR must personally sign and date

Participant/LAR
signature

Participant/LAR
name (Print)

LAR relationship to participant

information (data about myself/the participant); and (3) to state that I have received a signed and dated copy

| participant | | |
|---|---|---|
| Witness signature (if required) | | |
| Witness for non-English speaking participant: I declare that I am fluent in both English and in the participant's (or LAR's) language, and I confirm that the consent discussion was appropriately interpreted for the participant (or LAR). | | |
| Other: I confirm that the consent discussion occurred, and that the participant agreed to participate in this study by signing this form, making his/her mark, or verbally agreeing. | | |
| Name of witness: | | |
| Signature of witness: | | Date: |
| (The name of the witness must | t be documented in the EMR.) | |
| Interpreter (if required) | 1 | |
| Name of interpreter (if p | oresent): | |
| ID number (if phone into | erpreter): | |
| (The interpreter's name or ID r | number must be documented in the EM | MR.) |

The participant/Legally Authorized Representative must be provided with a signed copy of this form.



Memorial Sloan Kettering Cancer Center IRB Number: 21-442 A(5)
Approval date: 02-Aug-2023

# **Participant Assent for Clinical Research**

Assent is required for a minor age 7 to 17 and for a participant with mildly impaired decision-making capacity.

| Consenting Professional Must Personally Sign and Date | |
|---|---|
| Consenting Professional's Statement | |
| I have explained the study to the participant in age-appropriate terms and he/she agreed to take part in the study. He/she should sign and date below in the participant section. I have given a copy of this form to the participant and his/her Legally Authorized Representative (LAR). | |
| ☐ Check the box if the participant verbally agreed to take part but declined to sign or is unable to sign. | |
| Signature of | Date: |
| consenting<br>professional<br>obtaining assent | |
| Consenting professional name (printed) | |
| Participant Should Personally Sign and Date | |
| Participant's Statement | |
| I have read this consent or it was explained to me. All my questions have been answered. | |
| I agree to be in this research study. | |
| Participant<br>signature | Date: |

This form must be accompanied by an IRB-approved consent form signed by a Legally Authorized Representative.

